CLINICAL TRIAL: NCT03060668
Title: Optimized Caloric-proteic Nutrition in Critically Ill Patients: Impact on Short and Long-term Outcomes
Brief Title: Optimized Caloric-proteic Nutrition in Critically Ill Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Sao Domingos (Other)
Responsible Party: Principal Investigator, José Raimundo Araujo de Azevedo, PhD, Hospital Sao Domingos
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HSaoDomingos
Record Dates: First submitted 2017-02-11; First posted 2017-02-23 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2017-02

CONDITIONS: Critically Ill
Keywords: Critical Illness; Indirect Calorimetry; Dietary Proteins
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Caloric needs will be determined by indirect calorimetry. Patients in this group will receive 2.0 to 2.2 grams/kg/day of protein.
  Nutritional therapy will be initiated in the first 24 hours after admission.
  Nutritional formula will be Peptamen Intense (1.0 kcal/ml, 93 g/L protein (Nestle Health Care).
  Interventions: Other: Peptamen intense
- Control Group (Active Comparator): Patients in this group will receive 25 Kcal/kg/day and 1.4 to 1.5 grams/kg/day of protein.
  Nutritional formula in this group will be Novasource senior (Nestle Health Care).
  Nutritional therapy will be initiated in the first 24 hours after admission.
  Interventions: Other: Novasource senior

INTERVENTIONS:
Other: Peptamen intense — Study group will receive a nutritional formula containing 1.0 kcal/ml and 93 g/L of protein
  Arms: Study Group
Other: Novasource senior — Control group will receive a nutritional formula containing 1.2 kcal/ml and 65 g/L of protein
  Arms: Control Group

SUMMARY:
In this prospective randomized controlled trial the investigators intend to compare the use of a nutritional therapy based on caloric intake determined by indirect calorimetry and a high protein intake (2.0 to 2.2 g/kg/day) with a nutritional regimen based on 25 Kcal/kg/day and protein intake usually recommended to critically ill patients (1.4 to 1.5 grams/kg/day).

DETAILED DESCRIPTION:
OBJECTIVES

To evaluate the effect of nutritional therapy with caloric intake determined by indirect calorimetry and high protein intake (2.0 to 2.2 g/kg/day) compared to nutritional therapy with 25 kcal/kg/day and 1.4 to 1, 5 g/kg/day of protein on short-term outcomes and physical component (PCS) of quality of life after 3 and 6 months of randomization in severe ICU patients.

The primary objective will be the evaluation of the physical component summary (PCS) of SF-36 (Short Form 36), a questionnaire used to evaluate quality of life, validated for the Brazilian population. Patients will be assessed at least 3 and 6 months after randomization.

Secondary objectives: Measurement of handgrip strength measured on the 7th and 14th day of the study and on discharge from the ICU, ICU mortality, hospital mortality, mechanical ventilation time and length of stay in the ICU.

METHODS

The study will include patients over 18 years of age, not pregnant, submitted to mechanical ventilation, whose expectation of stay in the ICU is greater than 3 days.

The sample size was calculated based on the following parameters: patient population under mechanical ventilation, 528, 15% relative risk reduction in the evaluation parameter of the SF-36 tool, Level of significance (α) of 5%, test power of 80%, thus the number of individuals to be sampled will be 294, i.e., two groups of 147 patients. A computer-generated list for randomization and sequentially numbered opaque sealed envelopes is used. The level of significance to reject the null hypothesis will be 5%, that is, a value of p <0.05 will be considered as statistically significant.

Informed consent was obtained from the patient or a next of kin.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill patients Mechanically ventilated Expected length in the ICU > 3 days

Exclusion Criteria:

* Pregnancy Requirement for inspired oxygen (FIO2) > 0.60 High output bronchopleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
PCS of SF-36 | 6 months after randomization
  Physical component summary of Short Form 36

SECONDARY OUTCOMES:
Handgrip strength | 7th, 14th after admission and up to 30 days
  Measured using a calibrated dynamometer
ICU mortality | Up to 30 days
  ICU outcome
Hospital mortality | Up to 6 months
  Hospital outcome

CONTACTS AND LOCATIONS:
Overall Officials: JOSE R AZEVEDO, PhD, Principal Investigator — Hospital Sao Domingos
Locations (1):
- Hospital Sao Domingos, São Luís, Maranhão, Brazil

IPD SHARING:
Plan to Share IPD: No